CLINICAL TRIAL: NCT00625053
Title: Abdominal Midline Incisional Hernia Repair and Functional Outcome: Randomized Controlled Trial to Compare Open and Laparoscopic Surgical
Brief Title: Functional Outcome After Incisional Hernia Repair: Open Versus Laparoscopic Repair
Acronym: GINCISHERNIA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Ihsan INAN M.D., Geneva University Hospital, Department of Surgery, Visceral Surgery Division
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-293
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Hernia, Ventral; Body Image; Respiratory Function Tests; Quality of Life; Laparoscopy
Keywords: Neuroticism; Hernia, ventral; Laparoscopy; Quality of life
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Laparoscopic repair
  Interventions: Procedure: Laparoscopic repair
- 2 (Active Comparator): Open repair
  Interventions: Procedure: Open midline incisional hernia repair

INTERVENTIONS:
Procedure: Laparoscopic repair — Complete adhesiolysis between viscera and abdominal wall, complete dissection of round ligament and subumbilical fatty tissue to expose the posterior fascia at least 5 cm further than the cranial and caudal limits of the fascial defect or the original incision. Overlap of minimum 5 cm is calculated and mesh inserted in the abdominal cavity through 12mm optical trocar. Fixation of a antiadhesive composite mesh with helicoidal pins with maximum 15mm interval, double crown technique. No pressure decrease maneuver is done during mesh fixation or at another time during the operation. No transparietal suture fixation. No fascial closure.
  Other Names: TIP
  Arms: 1
Procedure: Open midline incisional hernia repair — * Underlay retromuscular repair: Medial border of the anterior fascia opened, posterior aspect of rectus muscle dissected to reach lateral border of rectus sheet, bilaterally. Peritoneum and posterior rectus fascia closed with absorbable running suture. Polyester or light-weight polypropylene mesh is cut to fit the reconstructed area, to have 3cm overlap on caudal and cranial defect limits. Mesh is fixed by absorbable sutures. Anterior fascia is closed with absorbable running suture. Components separation upon need.
  * Intraperitoneal onlay repair: Mesh is inserted intraperitoneally and fixed by a complete running suture (optional fixation with helicoidal pins or stapler). Fascial defect is closed with interrupted or running absorbable suture. Components separation upon need.
  Other Names: Stoppa-Rives
  Arms: 2

SUMMARY:
Background: Midline incisional hernia is reported from 0,5 to 11% after abdominal operations. Primary repair without mesh reinforcement is almost abandoned because of high recurrence rates (24 to 46%). Use of prosthetic mesh in incisional hernia repair lowered the recurrence rates under 10%. Recurrence rate alone is not the main quality criterion for incisional hernia repair anymore. Large series and meta-analyses confirmed the value of laparoscopic repair as at least equal if not better compared with open repair. Discomfort, pain, diminished quality of life and body image alteration influences functional well being. No baseline information exists in any of these fields treating pre- or post-operative phases in patients with incisional hernia. Respiratory functions and medico-economic evaluation are other rarely investigated fields that we consider in our trial. The objective of this study is to analyse the functional outcome status of patients after laparoscopic incisional hernia repair compared to open repair.

Methods: A randomized controlled non-blinded clinical trial is designed to compare laparoscopic incisional hernia mesh repair with open repair on post operative pain, health related quality of life outcomes, body image and cosmetic measurements, respiratory functions, recurrence rates, and cost. Volunteers will be recruited in Geneva University Hospital, department of surgery, visceral surgery unit. Eligibility criteria is male patient aged over 18 years, with reducible incisional hernia who are candidates for elective surgery and medically fit for general anesthesia.30 patients will be enrolled for each group. Follow-up will take place at 10th, 30th days as well as 3 12 and 24 post operative months by questionnaires and by clinical exam by independent expert. An overall cost-analysis will be realized. Patient enrollment in the study will start in April 2008 and estimated to end in september 2009.

DETAILED DESCRIPTION:
Midline incisional hernia is reported from 0,5 to 11% after abdominal operations. Discomfort, pain, body image alteration and diminished quality of life influences functional well being. Alteration in pulmonary function, risk of visceral incarceration or cutaneous complications are potential medical complications. Primary repair without mesh reinforcement is almost abandoned because of high recurrence rates (24 to 46%). Recurrence rate with prosthetic repair in published series vary from 4% to 29%. Different techniques for mesh placement and variety of mesh and fixation material explains this wide range of recurrence rate nevertheless, large series with standardized techniques report less than 4% of recurrence rates.

Laparoscopic repair for incisional hernia is first published in 1993. Following reported large personal series in recent years and evolution of adapted materiel, this technique gained popularity.

The main difference between open and laparoscopic techniques is the reconstruction of the abdominal wall. In all open techniques, abdominal wall is reconstructed (hernia edges brought together) with reinforcement of the abdominal wall by a mesh inserted onlay, sublay or inlay. In laparoscopic repair, the fascial defect is left in-situ but reinforced with a mesh, overlapping largely the edges of hernia.

Advocated advantages of laparoscopy are: less abdominal wall dissection (less surgical complications), tension-free mesh repair (no suturing), less postoperative pain, less respiratory complications, shorter hospital stay, faster return to professional activity. Disadvantages attributed to laparoscopic repair are the steep learning curve, high material cost, longer operation times and rare but serious complications.

Large series and meta analyses confirmed the value of laparoscopic repair as at least equal if not better compared with open repair. Most of the trials are focused on recurrence, complication rate, hospital stay and sick leave. Only recently, quality of life and pain started to be evaluated. No valuable data exists on chronic pain or persistent neuralgia, body image, cosmesis or neuroticism neither after open nor the laparoscopic repair.

Chronic pain or persistent neuralgia has been recognized as a complication after inguinal hernia repair but was reported in the 1980s as a rare and infrequent condition. Studies from the mid 1990s have reported a higher frequency, with up to 50% of patients reporting pain after hernia repair more than 1 year after surgery. Chronic pain after hernia repair can be disabling, with considerable impact on quality of life. The natural history of postoperative pain, including its prevalence, etiology, duration, associated disability and it's social and economical impact remain undefined.

We know from our experience in inguinal hernia that chronic pain needs to be investigated scrupulously to be identified. 20 to 27% chronic pain is associated to open repair in series without specific questionnaires. Overall frequency of chronic pain is higher in studies with specific measurements, where pain is the primary outcome of interest. Preoperative psychological state of patient (depression, dependencies, drug consumption etc.) or history of chronic pain with previous surgery or accident may be a predicting factor.

The definition of "chronic pain" by the International Association of the Study of Pain is "pain lasting for 3 months or more". There is no a consensus on neither in the definition, nor the severity grades of CSPOP in the literature. In our study chronic pain is defined as a minimal score > 4 using the quadruple visual analogue scale (VASQ) 3 months after procedure.

Somatic, and neuropathic chronic pain syndromes are described. Neuropathic pain usually develops in the sensory distribution of an injured nerve. Chronic residual neuralgia occurs as a result of surgical handing of sensory nerves. The nerve trauma can be due to partial or complete division, stretching, contusion, crushing, electrical damage, or sutures compression. Secondary nerve damage can occur due to irritation or compression by an adjacent inflammatory process such as granuloma. Neuropathic pain described as pulling, tugging, tearing, throbbing, stabbing, shooting, numbing, and dull. The onset of neuropathic pain is often delayed, occurring after a latent period of days to weeks. Pain is often aggravated by ambulation and sexual intercourse. Once chronic pain is installed, it does not change without a radical treatment. Preoperative psychological state of patient (Depression, dependencies, drug consumption etc.) or history of chronic pain with previous surgery or accident may be a predicting factor.

The definition of ''Body image'' is given as person's perception of, satisfaction with, and attitudes toward his or her body in general and to particular areas of the body. Little is known about the subjective feelings and cosmetic consequences of scarring in patients who undergo either conventional or laparoscopic abdominal surgery. Few data has been reported about body image in patients with cancer, particular after mutilating operations such as mastectomy. Three papers on ileocolectomy, proctectomy and live donor nephrectomy are published by Dutch groups, comparing laparoscopy and laparotomy. Body image in presence of an incisional hernia is certainly degraded before the surgery, unfortunately no baseline data exists to date. Therefore, an hypothetic, relative, significant improvement in body image by laparoscopic treatment compared to open repair needs to be evaluated.

The standard open technique in our institution has two declinations, the first technique is retromuscular sublay and the second, open onlay mesh repair. In both techniques the fascial defect is closed by suture repair with mesh reinforcement. Superiority of one of these techniques compared to another is not proved, properly done, both achieve low recurrence rates. Laparoscopic technique needs to meet widely accepted good-practice principles: complete adhesiolysis between abdominal wall and viscera, use of specific bilayer mesh (non adherent on the visceral surface), coverage of totality of the previous scar length with at least 5cm overlap, adequate fixation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 18 years or older
* Diagnosis of reducible incisional hernias up to 200 cm²
* Medically fit for general anesthesia
* Comprehension and use of French language
* Installed in the geographical region without foreseeable move for two years

Exclusion Criteria:

* Incarcerated hernia
* Ongoing chronic pain syndrome, other than hernia origin
* Coagulation disorders, prophylactic or therapeutic anticoagulation, unable to stop platelet antiaggregation therapy 10 days before surgery
* American Society of Anesthesiology Class 4 and 5 patients
* Emergency surgery, peritonitis, bowel obstruction, strangulation, perforation
* Mentally ill patients
* Presence of local or systemic infection
* Life expectancy < 2 years
* Any cognitive impairment (Psychiatric disorder, Alzheimer's disease etc.)
* Morbid obesity (BMI over 40)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Does Laparoscopic repair generate better functional outcome compared to the open mesh repair. Functional outcome includes pain, quality of life, body image and cosmetic measurements. | Preoperative, 10, 30, 90, 365 and 730 postoperative days

SECONDARY OUTCOMES:
Respiratory function | Preoperative, 10, 90 and 365 postoperative days
Influence of neuroticism on overall outcome | Preoperative, 10, 30, 90, 365 and 730 postoperative days
Postoperative surgical and medical complications | Preoperative, 10, 30, 90, 365 and 730 postoperative days
Overall cost analysis | Two years after the operation
Recurrence rate | Two years after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MOREL, Prof., Study Chair — Geneva University Hospital, Departement of Surgery, Visceral Surgery Division; Ihsan INAN, M.D., Study Director — Geneva University Hospital, Departement of Surgery, Visceral Surgery Division
Locations (1):
- Geneva University Hospital, Department of Surgery, Visceral Surgery Division, Geneva, Switzerland